CLINICAL TRIAL: NCT03397134
Title: A Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Monotherapy, 12-Week Study to Evaluate the Efficacy and Safety of 2 Fixed Doses of MIN-101 in Adult Patients With Negative Symptoms of Schizophrenia, Followed by a 40-Week Open-Label Extension
Brief Title: Study to Evaluate Efficacy and Safety of Roluperidone (MIN-101) in Adult Patients With Negative Symptoms of Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Minerva Neurosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MIN-101C07
Record Dates: First submitted 2017-12-29; First posted 2018-01-11 (Actual); Results first posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Negative Symptoms of Schizophrenia
MeSH Terms: interventions — roluperidone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Roluperidone 64 mg (Experimental): Roluperidone 64 mg for entire study
  Interventions: Drug: Roluperidone 64 mg
- Roluperidone 32 mg (Experimental): Roluperidone mg for entire study
  Interventions: Drug: Roluperidone 32 mg
- Placebo-1 (Placebo Comparator): Placebo for 12 weeks followed by Roluperidone 64 mg during open-label extension
  Interventions: Drug: Placebo Oral Tablet; Drug: Roluperidone 64 mg
- Placebo-2 (Placebo Comparator): Placebo for 12 weeks followed by Roluperidone 32 mg during open-label extension
  Interventions: Drug: Placebo Oral Tablet; Drug: Roluperidone 32 mg

INTERVENTIONS:
Drug: Placebo Oral Tablet — Placebo administered as a single dose once daily
  Arms: Placebo-1; Placebo-2
Drug: Roluperidone 32 mg — Roluperidone administered as a single dose once daily
  Arms: Placebo-2; Roluperidone 32 mg
Drug: Roluperidone 64 mg — Roluperidone administered as a single dose once daily
  Arms: Placebo-1; Roluperidone 64 mg

SUMMARY:
MIN-101C07 is a multicenter, multinational, randomized, double-blind, placebo-controlled, parallel-group study to evaluate the efficacy and safety of roluperidone in adult schizophrenia patients.The primary objective is to evaluate the efficacy of 2 fixed doses of roluperidone compared to placebo in improving the negative symptoms of schizophrenia over 12 weeks of double-blind treatment as measured by the change in Positive and Negative Syndrome Scale (PANSS) Marder negative symptoms factor score (NSFS) over 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patient and patient's legal representative, if applicable, provided informed consent prior to the initiation of any study related procedures, and the patient is judged by the investigator as being capable of understanding the study requirements.
* Male or female patient, 18 to 55 years of age, inclusive, and body mass index (BMI) < 35 kg/m(2) at Screening.
* Patient meets the diagnostic criteria for schizophrenia as defined in the Diagnostic and Statistical Manual of Mental Disorders (DSM-5), as established by a full psychiatric interview in conjunction with the Mini International Neuropsychiatric Interview.
* Has a reliable caregiver or family member or health care personnel who can provide information towards assessment and support the patient in terms of compliance with the protocol. The caregiver must have contacts with the patient daily for at least 1 hour each time and is not expected to change during the trial.
* Documented diagnosis of schizophrenia for at least 1 year before screening into the trial.
* Patient is stable in terms of positive and negative symptoms of schizophrenia over the last 6 months according to his or her treating psychiatrist and based on documentation in the clinical chart.
* Patient is currently an outpatient and has not been hospitalized for the last 6 months for acute exacerbation or symptoms worsening. Patients hospitalized during the last 6 months for social reasons or are currently hospitalized for social reasons can be included only with Sponsor's Responsible Medical Officer's approval, and the social reasons must be documented in the electronic case report form (eCRF).
* Patient with a score of > 20 on the PANSS negative subscore (the original PANSS scale [ Sum of N1+N2+N3+N4+N5+N6+N7]) at Screening (Visit 1) and Baseline (Visit 3) AND < 4 points absolute difference between 2 visits.
* Patients can be on any psychotropic before the trial if the psychotropics can be discontinued at the beginning of the washout phase without risking the patient's clinical status or safety.
* No history of violence against self or others during the last 1 year.
* Female patient who are not of childbearing potential, defined as women who are postmenopausal (defined as spontaneous amenorrhoea for at least 1 year or spontaneous amenorrhoea for at least 6 months confirmed by follicle stimulating hormone result of ≥ 40 IU/mL) or permanently sterilized (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy).
* Female patient, if of childbearing potential, must test negative for pregnancy and must be using a double barrier contraceptive method.
* Patient must be extensive metabolizers for cytochrome P450 (CYP2D6), defined as a subject that has at least one functional allel (e.g., *1 or *2), as determined by study-specific genotyping test before the first drug dose is administered.
* Patient and the caregiver are considered by the investigator to be reliable and likely to cooperate with the assessment procedures.

Exclusion Criteria:

* Current major depressive disorder, bipolar disorder, panic disorder, obsessive compulsive disorder, or intellectual disability (intellectual developmental disorder diagnosed by age 14).
* Patient with PANSS item score of > 4 on: P4 excitement/hyperactivity, P6 suspiciousness/persecution, P7 hostility, G8 uncooperativeness, G14 poor impulse control.
* A Calgary Depression Scale for Schizophrenia (CDSS) total score > 6.
* A score of ≥ 2 on any 2 items 1, 2, or 3, or a score of ≥ 3 on item 4 of the Barnes Akathisia Rating Scale (BARS).
* Patient's condition is due to direct psychological effects of a substance (e.g., a drug of abuse, or medication) or a general medical condition.
* Has a current or recent history of serious suicidal behavior within the past 1 year.
* Patient has a history of substance use disorder within 3 months of the Screening visit (excluding caffeine and cigarette smoking).
* Positive urine drug screen for drugs of abuse (cocaine, methadone, amphetamines, cannabinoids, opiates, benzodiazepines, and barbiturates), tricyclic antidepressants (TCA), and alcohol (except for prescription benzodiazepines).
* Patient who cannot be discontinued from psychotropics other than those allowed.
* Patient who received clozapine within 6 months of the Screening visit.
* Patient receiving treatment with long-acting or depot antipsychotic medication unless his/her next scheduled dose will occur during the protocol Screening period and can be omitted to allow for sufficient washout before receiving the study drug.
* Patient with a history of significant other major or unstable neurological, neurosurgical (e.g., head trauma), metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, or urological disorder.
* Patient with a history of seizures (patient with a history of a single childhood febrile seizure may be enrolled in this study).
* Patient who has had electroconvulsive therapy (ECT), vagal nerve stimulation (VNS), or repetitive trans-cranial magnetic stimulation (r-TMS) within the 6 months prior to the Screening visit or who are scheduled for ECT, VNS, or r-TMS at any time during the study.
* Patient with clinically significant abnormalities in hematology, blood chemistry, ECG, or physical examination not resolved by the Baseline visit which according to Investigator can interfere with study participation.
* Current systemic infection (e.g., Hepatitis B, Hepatitis C, human immunodeficiency virus [HIV], tuberculosis). Patients with positive Hepatitis B core antibody test and negative Hepatitis B surface Antigen (HBsAg) may be included in the study if aminotransferase levels (alanine aminotransferase (ALT)/ serum glutamic pyruvic transaminase (SGPT) [ALT/SGPT] and aspartate aminotransferase (AST)/ serum glutamic oxaloacetic transaminase (SGOT) [AST/SGOT] do not exceed 2 times upper limit of normal (ULN).
* Patient who requires or may require concomitant treatment with any other medication likely to increase QT interval (e.g., paroxetine, fluoxetine, duloxetine, amiodarone).
* Patient who requires medication inhibiting CYP 2D6 or CYP 3A4.
* Patient with a clinically significant ECG abnormality that could be a safety issue in the study, including QT interval value corrected for heart rate using the Fridericia's formula (QTcF) > 430 msec for males and > 450 msec for females.
* Patient with a history of myocardial infarction based on medical history or ECG findings at Screening.
* Familial or personal history of long QT syndrome or with additional risk factors for Torsade de Pointes.
* Subjects whose safety laboratory results show hypokalemia, hypomagnesemia, hypocalcemia.
* Patients with unexplained syncope.
* Woman of child-bearing potential, or man, who are unwilling or unable to use accepted methods of birth control.
* Woman with a positive pregnancy test, is lactating, or is planning to become pregnant during the study.
* Patient who participated in another clinical study within 3 months prior to Screening, or received roluperidone previously, or has previously participated in > 2 clinical studies with experimental medication (previous participation in 3 clinical studies with experimental medication will require approval of the sponsor before eligibility is determined).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 515 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2020-05-26 (Actual); Study Completion 2021-02-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (39):
- United States (13):
  - Woodland Research Northwest, Rogers, Arkansas
  - ProScience Research Group, Culver City, California
  - Collaborative Neuroscience Network, LLC., Garden Grove, California
  - Synergy Clinical Center, National City, California
  - Collaborative Neuroscience Network, LLC., Torrance, California
  - Behavioral Clinical Research, Inc, North Miami, Florida
  - Research Centers of America, LLC, Oakland Park, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Uptown Research Institute LLC, Chicago, Illinois
  - Hassman Research Institute, LLC., Berlin, New Jersey
  - The Nathan Kline Institute for Psychiatric Research, Orangeburg, New York
  - InSite Clinical Research LLC, DeSoto, Texas
  - Pillar Clinical Research LLC, Richardson, Texas
- Bulgaria (7):
  - "State Psychiatric Hospital - Tserova Koria"; Department for Active Treatment of Severe Psychosis - male; Department for Active Treatment of Severe Psychosis - male, Tserova Koria, Veliko Tarnovo District
  - "Mental Health Center Prof. Dr. Ivan Temkov - Burgas" EOOD Department For Treatment of Emergency Psychiatry Conditions, Burgas
  - State Psychiatry Hospital - Lovech, Lovech
  - State Psychiatry Hospital "Sveti Ivan Rilski" Department of General Psychiatry for adults "closed type" - males; Department of General Psychiatry for adults "closed type" - females, Novi Iskar
  - 'Mental Health Center Plovdiv"-EOOD Department for treatment of acute female/male psychoses with endogenous, exogenous, organic psychotic disturbances of the personality, Plovdiv
  - Multiprofile Hospital for Active Treatment - Targovishte" AD Department of Psychiatry, Targovishte
  - "Mental Health Center - Vratsa" General Psychiatric Department, Vratsa
- Poland (3):
  - Samodzielny Publiczny Psychiatryczny zakład opieki zdrowotnej im Dr. Stanisława Deresza w Choroszczy, Choroszcz
  - Medical University of Gdańsk, Department of Psychiatry UCK, Gdansk
  - Klinika Psychiatryczna Inventiva, Tuszyn
- Ukraine (16):
  - Communal Institution "Dnipropetrovsk Regional Clinical Hospital n.a. I.I. Mechnikov," Regional Centre for Psychosomatic Disorders based on Psychoneurological Department, Dnipro
  - Ivano-Frankivsk National Medical University (IFNMU) - Regional Psycho-Neurological Hospital #3, Ivano-Frankivsk
  - Kharkiv Railway Clinical Hospital N°1 of Branche "Health Center" of the Public joint stock company "Ukrainian Railway," Psychiatry Department, Kharkiv
  - State Institution "Institute of Neurology, Psychiatry and Narcology of National Academy of Medical Science of Ukraine," Department of Emergency Psychiatry and Narcology, Kharkiv
  - State Institution "Institute of Neurology, Psychiatry and Narcology of National Academy of Medical Science of Ukraine," Department of Neuroses and Borderline Conditions, Kharkiv
  - State Institution "Institute of Neurology, Psychiatry and Narcology of National Academy of Medical Sciences of Ukraine," Department of Clinical, Social and Child Psychiatry, Kharkiv
  - Kyiv Regional Medical Incorporation "Psychiatry," Centre of Novel Treatment and Rehabilitation of Psychotic Disorders based on Department #29 and Department #30, Kyiv
  - Communal Institution of Lviv Regional Council "Lviv Regional Clinical Psychiatric Hospital," Department #20, Lviv
  - Communal Institution of Lviv Regional Council "Lviv Regional Clinical Psychiatry Hospital," General Psychiatric Mixed Department #25, Lviv
  - Odessa Regional Medical Centre of Mental Health, Dept. #6 (male), Dept. #12 (female), Odesa
  - Kyiv Regional Medical Incorporation "Psychiatry," Centre of Novel Treatment and Rehabilitation of Psychotic Disorders based on Department #29 and Department #30, Oleksandrivka
  - "Ukrainian medical stomatological academy," Chair of psychiatry, narcology and medical psychology based on Poltava Regional Clinical Psychiatric Hospital named after O.F. Maltsev, female acute general psych. dept. 5-b, male acute general psych. dept 2-a, Poltava
  - Communal Institution "Cherkasy Regional Psychiatric Hospital", Smila
  - Municipal Institution Kherson Regional Psychiatric Hospital of Regional Council, Stepanovka
  - Ternopil Regional Municipal Clinical Psychoneurological Hospital, Ternopil
  - Municipal Institution "Vinnytsya Regional Psychoneurological Hospital n.a. Acad. O.I. Yushchenko," Male Department No 14, Female Department No 15, Vinnytsia

REFERENCES:
- [Result] Davidson M, Saoud J, Staner C, Noel N, Werner S, Luthringer E, Walling D, Weiser M, Harvey PD, Strauss GP, Luthringer R. Efficacy and Safety of Roluperidone for the Treatment of Negative Symptoms of Schizophrenia. Schizophr Bull. 2022 May 7;48(3):609-619. doi: 10.1093/schbul/sbac013. PMID 35211743

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the double-blind period, 857 patients were screened in the study, and 515 patients were randomized to receive treatment, including 172 patients in the placebo group and 343 patients in the Roluperidone group. Two patients who failed to meet eligibility criteria during screening, were randomized prematurely to the 32 mg Roluperidone group but were discontinued prior to receiving any study drug. Therefore, the total number of participants started is 513.
Groups:
- Placebo in Double Blind to Roluperidone 32 mg in Open Label: Placebo administered in double-blind period of study then to Roluperidone 32 mg during open-label extension period of study.
  Placebo administered as a single dose once daily.
  Roluperidone 32 mg: Roluperidone administered as a single dose once daily.
- Placebo in Double Blind to Roluperidone 64 mg in Open Label: Placebo administered in double-blind period of study then to Roluperidone 64 mg during open-label extension period of study.
  Placebo administered as a single dose once daily.
  Roluperidone 64 mg: Roluperidone administered as a single dose once daily.
- Roluperidone 32 mg at Any Time: Roluperidone 32 mg for entire study.
  Roluperidone 32 mg: Roluperidone administered as a single dose once daily.
- Roluperidone 64 mg at Any Time: Roluperidone 64 mg for entire study.
  Roluperidone 64 mg: Roluperidone administered as a single dose once daily.
- Placebo in Double Blind: Placebo in double-blind period of study.
  Placebo Oral Tablet: Placebo administered as a single dose once daily.
Period: Double Blind
Arm/Group | Placebo in Double Blind to Roluperidone 32 mg in Open Label | Placebo in Double Blind to Roluperidone 64 mg in Open Label | Roluperidone 32 mg at Any Time | Roluperidone 64 mg at Any Time | Placebo in Double Blind
Started | 0 | 0 | 170 | 171 | 172
Completed | 0 | 0 | 107 | 104 | 122
Not Completed | 0 | 0 | 63 | 67 | 50
Period: Open-Label Extension
Arm/Group | Placebo in Double Blind to Roluperidone 32 mg in Open Label | Placebo in Double Blind to Roluperidone 64 mg in Open Label | Roluperidone 32 mg at Any Time | Roluperidone 64 mg at Any Time | Placebo in Double Blind
Started | 59 | 63 | 107 | 104 | 0
Completed | 35 | 36 | 72 | 59 | 0
Not Completed | 24 | 27 | 35 | 45 | 0
Period: Whole Study
Arm/Group | Placebo in Double Blind to Roluperidone 32 mg in Open Label | Placebo in Double Blind to Roluperidone 64 mg in Open Label | Roluperidone 32 mg at Any Time | Roluperidone 64 mg at Any Time | Placebo in Double Blind
Started (Patients who were initially randomized in the double-blind to Roluperidone 32 mg or Roluperidone 64 mg continued treatment with the same dose during the 40-week open-label treatment extension, while patients who were initially randomized to placebo crossed over to Roluperidone 32 mg or Roluperidone 64 mg in a 1:1 ratio. The entire study included the double-blind and open-label periods from Baseline to Week 54, referred to as the "whole study period".) | 0 | 0 | 229 | 234 | 50
Completed | 0 | 0 | 107 | 95 | 0
Not Completed | 0 | 0 | 122 | 139 | 50

BASELINE CHARACTERISTICS:
Population: Patients who Started Treatment.
Groups:
- Roluperidone 64 mg: Roluperidone 64 mg for the double-blind period.
  Roluperidone 64 mg: Roluperidone administered as a single dose once daily.
- Roluperidone 32 mg: Roluperidone 32 mg for the double-blind period.
  Roluperidone 32 mg: Roluperidone administered as a single dose once daily.
- Placebo: Placebo for the double-blind period.
  Placebo Oral Tablet: Placebo administered as a single dose once daily.
- Total: Total of all reporting groups
Arm/Group | Roluperidone 64 mg | Roluperidone 32 mg | Placebo | Total
Number analyzed (Participants) | 171 | 170 | 172 | 513
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (9.3) | 41 (9.4) | 41 (8.7) | 41 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 64 | 66 | 198
  Male | 103 | 106 | 106 | 315
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 3 | 12
  Not Hispanic or Latino | 167 | 165 | 169 | 501
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 0 | 3
  Black or African American | 18 | 19 | 20 | 57
  White | 151 | 147 | 152 | 450
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 27 | 27 | 81
  Bulgaria | 36 | 37 | 40 | 113
  Georgia | 5 | 5 | 2 | 12
  Israel | 0 | 4 | 2 | 6
  Moldova | 6 | 8 | 5 | 19
  Poland | 6 | 5 | 8 | 19
  Romania | 19 | 18 | 13 | 50
  Ukraine | 72 | 66 | 75 | 213

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in PANSS Marder Negative Symptoms Factor Score (NSFS)
Description: The Marder negative symptoms factor score (NSFS) derived from the complete Positive and Negative Syndrome Scale (PANSS) has been the most frequently used scale in schizophrenia clinical studies focusing on negative symptoms The PANSS measures comprehensive psychiatric symptoms, including positive, negative, and general symptoms. The full PANSS rates the patient on 30 different symptoms from 1 (absent) to 7 (extreme) based on an interview as well as reports of family members or primary care hospital workers. The NSFS consists of the sum of the negative symptom PANSS items N1, N2, N3, N4, N6, G7, and G16 (minimum score = 7; maximum score = 49). Higher scores indicate more severe symptoms.
Time Frame: Baseline, Week 2, Week 4, Week 8, and Week 12
Population: mITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Roluperidone 32 mg | Roluperidone 64 mg | Placebo
Number analyzed (Participants) | 167 | 162 | 167
score on a scale
  Baseline | 25.2 (3.43) | 25.3 (3.26) | 24.3 (3.01)
  Change from Baseline to Week 2 | -1.2 (2.22) | -1.7 (2.47) | -1.2 (2.46)
  Change from Baseline to Week 4 | -2.6 (2.57) | -2.8 (2.92) | -1.8 (2.99)
  Change from Baseline to Week 8 | -3.4 (3.49) | -3.8 (3.32) | -2.8 (3.44)
  Change from Baseline to Week 12 | -3.7 (3.20) | -4.5 (3.85) | -3.5 (3.97)
Statistical Analysis 1: Comparison: Roluperidone 64 mg vs Placebo; To evaluate the efficacy of 2 fixed doses (32 mg and 64 mg) of MIN-101 compared to placebo in improving the negative symptoms of schizophrenia as measured by the change from Baseline in the PANSS Marder negative symptoms factor score (NSFS) over 12 weeks of double-blind treatment. Approximation 501 eligible patients will be randomized in a 2:2:1:1 ratio at baseline to 1 of 4 treatment arms; Test type: Superiority — All statistical tests will be 2-sided hypothesis tests performed at the 5% level of significance. All confidence intervals will be 2-sided 95% confidence intervals; p = 0.043, Mixed Models Analysis — The p-values must be ≤0.025 to allow for rejecting the null hypothesis for the representative dose; The Kenward-Roger approximation will be used to estimate denominator degrees of freedom

2. Secondary Outcome: Change From Baseline to Week 12 in Personal and Social Performance (PSP)
Description: The PSP scale is a validated clinician-rated scale that measures personal and social functioning in 4 domains: socially useful activities (eg, work and study), personal and social relationships, self care, and disturbing and aggressive behaviors. It is a reliable, quick measure of personal and social functioning of patients with schizophrenia and can be used on patients in the acute and stable stage. PSP is a 100-point scale, divided into 10 equal intervals. The score is based on the assessment of a patient's performance in the 4 domains. Lower scores of 1 to 30 reflected poor functioning that the patient required intensive support or supervision; scores of 31 to 60 reflected varying degrees of disability; and scores of 71 to 100 reflected absence of disability or only mild difficulties.
Time Frame: Baseline, Week 4, Week 8, and Week 12
Population: mITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Roluperidone 32 mg | Roluperidone 64 mg | Placebo
Number analyzed (Participants) | 167 | 162 | 167
score on a scale
  Baseline | 52.7 (12.28) | 53.0 (10.60) | 52.9 (11.02)
  Change from Baseline to Week 4 | 1.6 (6.10) | 3.2 (6.30) | 1.2 (5.92)
  Change from Baseline to Week 8 | 3.6 (7.09) | 5.0 (6.76) | 3.1 (7.82)
  hange from Baseline to Week 12 | 4.6 (7.98) | 6.2 (8.67) | 4.2 (7.48)
Statistical Analysis 1: Comparison: Roluperidone 64 mg vs Placebo; The PSP involves four subscale domains: (a) socially useful activities, (b) personal and social relationships, (c) self-care, and (d) disturbing and aggressive behaviors. After each of these four areas is scored on an anchored Likert-type scale (0-5), raters are instructed to select a 10-point range within a 100-point scale, guided by the area scores assigned during assessment; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.016, Mixed Models Analysis — The p-values must be ≤0.025 to allow for rejecting the null hypothesis for the representative dose; The Kenward-Roger approximation will be used to estimate denominator degrees of freedom

3. Secondary Outcome: Change From Baseline to Week 12 in Clinical Global Impression of Severity (CGI-S)
Description: The Clinical Global Impression of Severity (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis: "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?" which is rated on the following seven-point scale: 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients
Time Frame: Baseline, Week 2, Week 4, Week 8, and Week 12
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo: Placebo for the double-blind period of study.
  Placebo Oral Tablet: Placebo administered as a single dose once daily.
Arm/Group | Roluperidone 32 mg | Roluperidone 64 mg | Placebo
Number analyzed (Participants) | 170 | 171 | 172
score on a scale
  Baseline | 4.0 (0.62) | 4.0 (0.61) | 4.0 (0.58)
  Change from Baseline to Week 2 | -0.1 (0.44) | -0.1 (0.54) | -0.1 (0.50)
  Change from Baseline to Week 4 | -0.2 (0.49) | -0.3 (0.55) | -0.1 (0.44)
  Change from Baseline to Week 8 | -0.3 (0.61) | -0.4 (0.68) | -0.2 (0.60)
  Change from Baseline to Week 12 | -0.4 (0.68) | -0.4 (0.67) | -0.3 (0.63)

4. Secondary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Values (Whole Study Period; Safety Population)
Description: Laboratory abnormalities were determined using pre-defined normal ranges. Clinical laboratory values were considered potentially clinically significant (PCS) for select parameters of hematology, chemistry, and urinalysis. The number and percentage of patients experiencing PCS laboratory abnormalities post-baseline were summarized by treatment group.
Time Frame: Entire study (which includes double-blind and open-label periods) from Baseline to Week 54 (referred to as the "whole study period")
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Roluperidone 32 mg: Roluperidone 32 mg for entire study.
  Roluperidone 32 mg: Roluperidone administered as a single dose once daily.
Arm/Group | Roluperidone 32 mg | Roluperidone 64 mg | Placebo
Number analyzed (Participants) | 229 | 234 | 172
Participants
  Low potentially clinically significant laboratory values | 43 | 37 | 18
  High potentially clinically significant laboratory values | 51 | 48 | 21

5. Secondary Outcome: Number of Participants With Potentially Clinically Significant ECG Parameters (Whole Study Period; Safety Population)
Description: QTcF values were tabulated for their absolute values and tabulated relative to Baseline measurements in order to detect individual QTcF changes. The number and percentage of patients who met criteria for potentially clinically significant (PCS) values were summarized.
Time Frame: as for outcome 4
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Roluperidone 32 mg | Roluperidone 64 mg | Placebo
Number analyzed (Participants) | 229 | 234 | 172
Participants
  Highest absolute QTcF interval > 450 -480 msec | 10 | 24 | 1
  Highest absolute QTcF interval > 480 -500 msec | 0 | 2 | 0
  Highest absolute QTcF interval > 500 msec | 0 | 2 | 0

6. Secondary Outcome: Number of Participants With Potentially Clinically Significant Vital Signs (Whole Study Period; Safety Population)
Description: The number and percentage of patients with any potentially clinically significant (PCS) vital sign (systolic blood pressure, diastolic blood pressure, heart rate/pulse rate, temperature) occurring post-Baseline were summarized.
Time Frame: as for outcome 4
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Placebo in double-blind period of study.
  Placebo Oral Tablet: Placebo administered as a single dose once daily.
Arm/Group | Roluperidone 32 mg | Roluperidone 64 mg | Placebo
Number analyzed (Participants) | 229 | 234 | 172
Participants | 37 | 28 | 20

7. Secondary Outcome: Safety Assessment - Abnormal Involuntary Movement Scale (AIMS)
Description: AIMS is rating scale that was designed to measure tardive dyskinesia (TD). For the scoring, the AIMS scale has 14 items. The first 10 items (under categories of Facial and Oral Movements, Extremity Movements, Trunk Movements, and Global Judgements) are rated from 0 (none) to 4 (severe); the remaining 4 items (Dental Status) are rated "yes" and "no" and not counted. The analysis is limited to items 1 to 10, with each rated from 0 to 4. The total score is the sum of all 10 items and with values ranging from 0 to 40. For the analysis, the observed composite movement (total) score will be summarized by treatment group and study visit. Higher scores imply worse outcome.
Time Frame: Study Baseline Day -1, Active Baseline last assessment on placebo at Week 12, as appropriate, Weeks 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 54. Active Baseline=last assessment before receiving Roluperidone.
Population: Safety Population
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo in DB to Roluperidone 32 mg in OL Extension: Placebo administered in double-blind period of study then to Roluperidone 32 mg during open-label extension period of study.
  Placebo administered as a single dose once daily.
  Roluperidone 32 mg: Roluperidone administered as a single dose once daily.
- Placebo in DB to Roluperidone 64 mg in OL Extension: Placebo administered in double-blind period of study then to Roluperidone 64 mg during open-label extension period of study.
  Placebo administered as a single dose once daily.
  Roluperidone 64 mg: Roluperidone administered as a single dose once daily.
Arm/Group | Placebo in DB to Roluperidone 32 mg in OL Extension | Placebo in DB to Roluperidone 64 mg in OL Extension | Roluperidone 32 mg at Any Time | Roluperidone 64 mg at Any Time
Number analyzed (Participants) | 86 | 86 | 170 | 171
score on a scale
  Study Baseline | 0.2 (1.23) | 0.1 (0.62) | 0.4 (1.40) | 0.3 (1.04)
  Active Baseline: number analyzed (Participants) | 59 | 63 | 107 | 104
  Active Baseline | 0.2 (1.45) | 0.1 (0.52) | 0.4 (1.20) | 0.3 (1.15)
  Week 16: number analyzed (Participants) | 51 | 54 | 103 | 97
  Week 16 | 0.2 (0.88) | 0.1 (0.56) | 0.5 (1.38) | 0.2 (1.18)
  Week 20: number analyzed (Participants) | 51 | 54 | 99 | 95
  Week 20 | 0.1 (0.50) | 0.1 (0.56) | 0.4 (1.60) | 0.2 (1.06)
  Week 24: number analyzed (Participants) | 50 | 51 | 92 | 81
  Week 24 | 0.1 (0.51) | 0.1 (0.57) | 0.4 (1.31) | 0.2 (1.37)
  Week 28: number analyzed (Participants) | 48 | 49 | 88 | 76
  Week 28 | 0.1 (0.52) | 0.1 (0.59) | 0.4 (1.30) | 0.2 (1.38)
  Week 32: number analyzed (Participants) | 42 | 47 | 88 | 74
  Week 32 | 0.1 (0.55) | 0.1 (0.60) | 0.4 (1.19) | 0.2 (1.45)
  Week 36: number analyzed (Participants) | 41 | 43 | 84 | 68
  Week 36 | 0.1 (0.69) | 0.1 (0.63) | 0.4 (1.29) | 0.2 (1.48)
  Week 40: number analyzed (Participants) | 40 | 42 | 80 | 67
  Week 40 | 0.1 (0.56) | 0.1 (0.63) | 0.3 (1.06) | 0.3 (1.53)
  Week 44: number analyzed (Participants) | 37 | 41 | 80 | 62
  Week 44 | 0.1 (0.33) | 0.0 (0.16) | 0.3 (1.17) | 0.1 (0.40)
  Week 48: number analyzed (Participants) | 37 | 38 | 74 | 61
  Week 48 | 0.1 (0.36) | 0.2 (0.59) | 0.4 (1.38) | 0.3 (1.57)
  Week 52: number analyzed (Participants) | 36 | 35 | 69 | 57
  Week 52 | 0.1 (0.33) | 0.0 (0.17) | 0.3 (1.31) | 0.3 (1.63)
  Week 54: number analyzed (Participants) | 35 | 34 | 71 | 57
  Week 54 | 0.1 (0.34) | 0.0 (0.17) | 0.5 (1.55) | 0.3 (1.63)

8. Secondary Outcome: Safety Assessments - Barnes Akathisia Rations Scale (BARS)
Description: The BARS is a multiple-choice questionnaire that clinicians used to provide an assessment of akathisia. The BARS scale has 3 items that are rated from 0 (absence/no distress) to 3 (most severe). The BARS rating scale is scored by summing the scales for Objective Akathisia, Subjective Awareness of Restlessness and Subjective Distress Related to Restlessness yielding a total score ranging from 0 to 9. The Total score, which has a possible range from 0-9, is reported. Higher scores imply worse outcome.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 8, and Week 12
Population: Safety Population
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Roluperidone 32 mg: Roluperidone 32 mg for the double-blind period.
  Roluperidone 32 mg: Roluperidone administered as a single dose once dail
Arm/Group | Roluperidone 32 mg | Roluperidone 64 mg | Placebo
Number analyzed (Participants) | 170 | 171 | 172
score on a scale
  Baseline | 0.1 (0.39) | 0.1 (0.42) | 0.1 (0.39)
  Week 1 | 0.1 (0.49) | 0.1 (0.39) | 0.1 (0.34)
  Week 2 | 0.2 (0.55) | 0.1 (0.47) | 0.1 (0.41)
  Week 3 | 0.1 (0.52) | 0.1 (0.43) | 0.1 (0.32)
  Week 4 | 0.1 (0.41) | 0.1 (0.41) | 0.1 (0.32)
  Week 8 | 0.1 (0.40) | 0.1 (0.44) | 0.0 (0.27)
  Week 12 | 0.1 (0.46) | 0.1 (0.37) | 0.0 (0.22)

9. Secondary Outcome: Safety Assessments -Simpson-Angus Scale (S-AS) Score
Description: The S-AS is an established reliable and valid rating scale that measures drug-induced extrapyramidal syndromes using 10 items rated from 0 = not present to 4 = extremely severe. It consisted of 1 item measuring gait (hypokinesia), 6 items measuring rigidity (arm dropping, shoulder shacking, elbow rigidity, wrist rigidity, leg pendulousness, and head dropping) and 3 items measuring glabella tap, tremor, and salivation. As such, the range of scores was 0 to 40, with increased scores indicating increased severity.
Time Frame: Study Baseline Day -1, Active Baseline last assessment on placebo at Week 12, as appropriate, Weeks 13, 14, 15, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 54. Active Baseline=last assessment before receiving Roluperidone.
Population: Safety Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo in DB to Roluperidone 32 mg in OL Extension | Placebo in DB to Roluperidone 64 mg in OL Extension | Roluperidone 32 mg at Any Time | Roluperidone 64 mg at Any Time
Number analyzed (Participants) | 86 | 86 | 170 | 171
score on a scale
  Study Baseline | 0.4 (0.80) | 0.5 (1.25) | 0.8 (2.18) | 0.6 (1.53)
  Active Baseline: number analyzed (Participants) | 59 | 63 | 107 | 104
  Active Baseline | 0.3 (0.83) | 0.1 (0.48) | 0.8 (2.10) | 0.5 (1.44)
  Week 13: number analyzed (Participants) | 54 | 61 | 97 | 94
  Week 13 | 0.2 (0.63) | 0.2 (0.60) | 0.8 (1.84) | 0.3 (1.04)
  Week 14: number analyzed (Participants) | 54 | 58 | 103 | 96
  Week 14 | 0.3 (0.81) | 0.2 (0.64) | 0.7 (1.77) | 0.4 (1.56)
  Week 15: number analyzed (Participants) | 53 | 59 | 105 | 97
  Week 15 | 0.2 (0.48) | 0.2 (0.64) | 0.7 (1.74) | 0.5 (1.61)
  Week 16: number analyzed (Participants) | 52 | 54 | 104 | 97
  Week 16 | 0.1 (0.34) | 0.1 (0.52) | 0.7 (1.68) | 0.5 (1.63)
  Week 20: number analyzed (Participants) | 51 | 54 | 99 | 95
  Week 20 | 0.1 (0.33) | 0.1 (0.52) | 0.6 (1.65) | 0.5 (1.64)
  Week 24: number analyzed (Participants) | 50 | 51 | 92 | 81
  Week 24 | 0.1 (0.40) | 0.1 (0.52) | 0.6 (1.56) | 0.5 (1.73)
  Week 28: number analyzed (Participants) | 48 | 49 | 88 | 76
  Week 28 | 0.2 (0.48) | 0.1 (0.53) | 0.7 (1.65) | 0.3 (1.66)
  Week 32: number analyzed (Participants) | 42 | 47 | 88 | 74
  Week 32 | 0.2 (0.49) | 0.1 (0.54) | 0.6 (1.60) | 0.4 (1.68)
  Week 36: number analyzed (Participants) | 41 | 43 | 84 | 68
  Week 36 | 0.2 (0.50) | 0.1 (0.54) | 0.6 (1.65) | 0.4 (1.70)
  Week 40: number analyzed (Participants) | 40 | 42 | 81 | 67
  Week 40 | 0.1 (0.30) | 0.1 (0.57) | 0.6 (1.36) | 0.4 (1.69)
  Week 44: number analyzed (Participants) | 37 | 41 | 80 | 62
  Week 44 | 0.3 (0.77) | 0.1 (0.35) | 0.6 (1.56) | 0.3 (0.82)
  Week 48: number analyzed (Participants) | 37 | 38 | 74 | 61
  Week 48 | 0.4 (1.52) | 0.1 (0.32) | 0.7 (1.69) | 0.5 (1.79)
  Week 52: number analyzed (Participants) | 36 | 35 | 69 | 57
  Week 52 | 0.1 (0.35) | 0.1 (0.34) | 0.5 (1.42) | 0.5 (1.84)
  Week 54: number analyzed (Participants) | 35 | 34 | 71 | 57
  Week 54 | 0.2 (0.49) | 0.2 (0.76) | 0.7 (1.75) | 0.5 (1.83)

10. Secondary Outcome: Safety Assessments - Sheehan Suicidality Tracking Scale (STS) Total Score
Description: Sheehan Suicidality Tracking Scale (STS) is a prospective rating scale that tracks treatment-emergent suicidal ideation and behaviors.
  Scoring: Each item is scored on a 5-point Likert scale from 0 (not at all) to 4 (extremely). Data from the STS can be analyzed as individual item scores, a subscore for suicidal ideation (sum of scores from items 2, 3, and 4, plus score from item 5 if ≤ 1), a subscore for suicidal behavior (sum of scores from items 6, 7, and 8, plus score from item 5 if > 1) and the total scale score (calculated by add scores from Questions 1a (only if 1b is coded YES), + 2 through 11 + [the highest of 12 or any row of 16] + [the highest of 14 or any row of 15] + 17 + 20.
  Analysis: The total scale score will be summarized by treatment group and study visit. Complete data will be presented in patient data listings by treatment group and visit. The total score is the sum of all 16 questions and with values ranging from 0 to 64. Higher scores imply worse outcome.
Time Frame: as for outcome 9
Population: Safety Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo in DB to Roluperidone 32 mg in OL Extension | Placebo in DB to Roluperidone 64 mg in OL Extension | Roluperidone 32 mg at Any Time | Roluperidone 64 mg at Any Time
Number analyzed (Participants) | 86 | 86 | 170 | 171
score on a scale
  Study Baseline: number analyzed (Participants) | 86 | 85 | 170 | 171
  Study Baseline | 0.0 (0.00) | 0.0 (0.15) | 0.0 (0.46) | 0.0 (0.08)
  Active Baseline: number analyzed (Participants) | 59 | 63 | 107 | 104
  Active Baseline | 0.0 (0.13) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.10)
  Week 12.1: number analyzed (Participants) | 58 | 62 | 106 | 104
  Week 12.1 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Week 12.2: number analyzed (Participants) | 59 | 63 | 105 | 102
  Week 12.2 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Week 13: number analyzed (Participants) | 54 | 61 | 98 | 95
  Week 13 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.10)
  Week 14: number analyzed (Participants) | 55 | 57 | 103 | 96
  Week 14 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Week 15: number analyzed (Participants) | 52 | 60 | 103 | 96
  Week 15 | 0.0 (0.14) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Week 16: number analyzed (Participants) | 53 | 55 | 103 | 97
  Week 16 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.10) | 0.0 (0.0)
  Week 20: number analyzed (Participants) | 51 | 53 | 100 | 94
  Week 20 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.41)
  Week 24: number analyzed (Participants) | 50 | 51 | 89 | 81
  Week 24 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Week 28: number analyzed (Participants) | 48 | 49 | 88 | 75
  Week 28 | 0.2 (1.44) | 0.0 (0.0) | 0.0 (0.11) | 0.0 (0.0)
  Week 32: number analyzed (Participants) | 41 | 47 | 88 | 74
  Week 32 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Week 36: number analyzed (Participants) | 41 | 43 | 83 | 68
  Week 36 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.11) | 0.0 (0.0)
  Week 40: number analyzed (Participants) | 38 | 43 | 82 | 67
  Week 40 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.11) | 0.0 (0.0)
  Week 44: number analyzed (Participants) | 37 | 41 | 80 | 62
  Week 44 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.22) | 0.0 (0.0)
  Week 48: number analyzed (Participants) | 37 | 38 | 75 | 61
  Week 48 | 0.1 (0.49) | 0.0 (0.0) | 0.0 (0.12) | 0.0 (0.38)
  Week 52: number analyzed (Participants) | 34 | 35 | 68 | 57
  Week 52 | 0.0 (0.17) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Week 54: number analyzed (Participants) | 34 | 34 | 71 | 59
  Week 54 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)

ADVERSE EVENTS:
Time Frame: Entire study (which includes double-blind and open-label periods) from Baseline to Week 54 (referred to as the "whole study period").
Description: Safety population=513 patients treated across the whole study period: 172 patients received at least 1 dose of placebo & 463 patients received at least 1 dose of roluperidone (including 229 patients who received 32 mg roluperidone & 234 patients who received 64 mg roluperidone). Of the 172 patients who received placebo during double blind, 122 patients continued into the open-label period. Of these 122 patients, 59 patients received 32 mg roluperidone & 63 patients received 64 mg roluperidone.
Groups:
- Placebo in Double Blind to Roluperidone 32 mg in Open Label: Placebo administered double blind Phase of Study then Roluperidone 32 mg during open label phase of study.
  Roluperidone 32 mg: Roluperidone administered as a single dose once daily
- Placebo in Double Blind to Roluperidone 64 mg in Open Label: Placebo administered double blind Phase of Study then Roluperidone 64 mg during open label phase of study.
  Roluperidone 64 mg: Roluperidone administered as a single dose once daily
- Roluperidone 32 mg at Any Time: Roluperidone 32 mg for entire study
  Roluperidone 32 mg: Roluperidone administered as a single dose once daily
- Roluperidone 64 mg at Any Time: Roluperidone 64 mg for entire study
  Roluperidone 64 mg: Roluperidone administered as a single dose once daily
- Placebo: Placebo
  Placebo Oral Tablet: Placebo administered as a single dose once daily
Arm/Group | Placebo in Double Blind to Roluperidone 32 mg in Open Label | Placebo in Double Blind to Roluperidone 64 mg in Open Label | Roluperidone 32 mg at Any Time | Roluperidone 64 mg at Any Time | Placebo
All-Cause Mortality (participants affected / at risk) | 0/59 | 1/63 | 2/229 | 1/234 | 0/172
Serious Adverse Events (participants affected / at risk) | 1/59 | 5/63 | 18/229 | 21/234 | 5/172
Other Adverse Events (participants affected / at risk) | 2/59 | 7/63 | 30/229 | 39/234 | 22/172
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo in Double Blind to Roluperidone 32 mg in Open Label (N=59) | Placebo in Double Blind to Roluperidone 64 mg in Open Label (N=63) | Roluperidone 32 mg at Any Time (N=229) | Roluperidone 64 mg at Any Time (N=234) | Placebo (N=172)
Schizophrenia (Psychiatric disorders) | 1 | 0 | 9 | 9 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 2 | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 2 | 0
Aggression (Psychiatric disorders) | 0 | 1 | 1 | 1 | 0
Psychotic symptom (Psychiatric disorders) | 0 | 0 | 1 | 1 | 3
Sleep Disorder (Psychiatric disorders) | 0 | 1 | 1 | 1 | 1
Completed suicide (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Hallucination, auditory (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Bartholinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Pneumonia viral (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo in Double Blind to Roluperidone 32 mg in Open Label (N=59) | Placebo in Double Blind to Roluperidone 64 mg in Open Label (N=63) | Roluperidone 32 mg at Any Time (N=229) | Roluperidone 64 mg at Any Time (N=234) | Placebo (N=172)
Insomnia (Psychiatric disorders) | 1 | 0 | 7 | 4 | 7
Schizophrenia (Psychiatric disorders) | 0 | 0 | 6 | 5 | 5
Agitation (Psychiatric disorders) | 0 | 0 | 4 | 4 | 2
Headache (Nervous system disorders) | 1 | 5 | 8 | 15 | 4
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 2 | 5 | 0
Asthenia (General disorders) | 0 | 1 | 3 | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/34/NCT03397134/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/34/NCT03397134/SAP_001.pdf